CLINICAL TRIAL: NCT03280992
Title: Community Acquired Sepsis Cohort
Acronym: CASC
Status: Terminated | Type: Observational
Why Stopped: Study not feasible in practise
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3024_CASC
Record Dates: First submitted 2017-08-18; First posted 2017-09-13 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Severe Septic Syndrome; Septic Shock
MeSH Terms: conditions — Toxemia; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to constitute a prospective cohort of all the patients presenting to the adult emergencies of the University Hospital Centre (CHU) of Rennes for a septic syndrome of community origin.

DETAILED DESCRIPTION:
Severe septic syndrome (SSG) and septic shock (CS) are two frequent and serious complications of infectious diseases. In this context, the optimization of the management of septic patients from their reception in the emergency services must be a priority. However there are no predictors of progression or severity in patients admitted to emergencies despite the recommendations emphasizing the need for screening and early therapeutic management. Many scores have been proposed for intensive care unit but they remain difficult to extrapolate to other services because they are very comprehensive and require information that is difficult to obtain for emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient hospitalized during the study period for community infectious diseases at the CHU of Rennes

Exclusion Criteria:

* Written objection from the patient to the computer processing of his data
* Pregnant women
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a community infectious diseases
Sampling Method: Non-Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Assessment of morbidity in patients with septic syndrome of community origin | Day 90
  Study of prognostic factors
Internal validity, severity score | Day 90
Internal validity, triage score by orientation nurses | Day 90
Study of the prognostic factors of patients with septic syndrome of community origin in terms of mortality | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France